CLINICAL TRIAL: NCT05354245
Title: Using a Complex Carbohydrate Mixture Added to a High-protein Diet to Steer Fermentation and Improve Metabolic, Gut and Brain Health
Brief Title: Using a Complex Carbohydrate Mixture to Steer Fermentation and Improve Metabolism in Adults With Overweight and Prediabetes (DISTAL)
Acronym: DISTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Carbohydrate Competence Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL80459.068.22
Record Dates: First submitted 2022-02-22; First posted 2022-04-29 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Insulin Resistance; Impaired Glucose Tolerance; PreDiabetes; Overweight and Obesity
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Prediabetic State; Overweight; Obesity | interventions — maltodextrin; Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibre mixture group (Experimental): Use of a fibre mixture (3 times daily, 5 grams per gift, total of 15 grams per day) during 12 weeks
  Interventions: Dietary Supplement: Fibre supplement (potato-pectin); Dietary Supplement: High-protein diet
- Placebo group (Placebo Comparator): Use of a placebo (maltodextrin, isocaloric manner, 3 times daily) during 12 weeks.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: High-protein diet

INTERVENTIONS:
Dietary Supplement: Fibre supplement (potato-pectin) — Fibre supplement
  Arms: Fibre mixture group
Dietary Supplement: Placebo — Maltodextrin
  Other Names: Maltodextrin
  Arms: Placebo group
Dietary Supplement: High-protein diet — High-protein diet

SUMMARY:
The purpose of this study is to investigate the effects of a fibre mixture added to a high-protein diet on metabolic, gut and brain health.

DETAILED DESCRIPTION:
The fibre mixture that will be investigated is hypothesized to improved metabolic, gut and brain health. It potentially increases insulin sensitivity, satiety, gut barrier function, improves food-reward related brain activity and decreases inflammation, gut permeability, and ectopic lipid accumulation, among other potential health effects.

The fibre mixture will be administrated during 12 weeks combined a high-protein diet. The placebo-controlled parallel design of the study allows for a placebo group to use maltodextrin combined with a high-protein diet for 12 weeks. The high-protein diet is known to increase satiety and might enhance the difference between the intervention and placebo groups in terms of outcome measurements. The potential health effects as described earlier will be investigated using different techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* Male/female
* BMI 28-40 kg/m2
* Impaired fasting glucose or glucose tolerance, determined using the following criteria (participant should meet at least one criteria):
* HbA1c 42-47 mmol/mol OR fasting glucose (>10h fasted) 5.6-6.9 mmol/l OR Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) >1.85

Exclusion Criteria:

* Diabetes mellitus (type 1 or 2)
* Cardiovascular disease (except hypertension (<160/100mmHg is allowed), pulmonary disease, kidney disease/failure, liver disease/failure
* Gastrointestinal disease or a history of abdominal surgery (except appendectomy and cholecystectomy)
* Diseases affecting glucose and/or lipid metabolism
* Malignancy (except non-invasive skin cancer)
* Auto-immune disease
* Major mental disorders
* Ongoing (infectious) disease or any disease with a life expectancy ≤5 years
* Substance abuse (nicotine abuse (including e-cigarettes) defined as >20 cigarettes per day; alcohol abuse defined as ≥8 drinks/week for females and ≥15 drinks/week for males(38); any drugs)
* A change in weight ≥3kg over the last 3 months or plans to lose weight or follow a hypocaloric diet during the study period
* Pre/pro/antibiotic use in the last 3 months or during the study
* Use of medication that influences glucose or fat metabolism and inflammation, such as:

  * Use of statins (stable use ≥3 months prior to and during study is allowed)
  * Use of antidepressants (stable use ≥3 months prior to and during study is allowed)
  * Use of specific anticoagulants
  * Use of medication known to interfere with study outcomes
  * Use of β-blockers
  * Chronic corticosteroid treatment (>7 consecutive days)
* Regular use of laxatives 3 months prior to the study or during study period
* Change in physical activity or diet during study period
* Intensive physical activity (>3h per week)
* Pregnancy
* Following a vegan or vegetarian diet; presence of food allergies, intolerances or diet restrictions interfering with the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | 12 weeks
  Change in peripheral insulin sensitivity between the two groups. Measured using a two-step hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
Insulin sensitivity (hepatic and adipose tissue) | 12 weeks
  Change in insulin sensitivity between the two groups. Measured using a two-step hyperinsulinemic-euglycemic clamp
Gut permeability | 12 weeks
  Difference in change between the groups. Measured using multisugar test
Inflammation | 12 weeks
  Difference in change between the groups. Measured using serum values.
Energy and substrate metabolism | 12 weeks
  Difference in change between the groups. Measured using serum values (circulating metabolites) and indirect calorimetry (energy harvest and expenditure)
Neurocognitive functioning | 12 weeks
  Difference in change between the groups. Measured using neurocognitive tests and functional Magnetic Resonance Imaging (fMRI).
  Neurocognitive functioning will be measured using the Cambridge Neuropsychological Test Automated Battery (CANTAB) (a combination of different digital tests) to assess response time in seconds and quality of delivered results. fMRI assesses food-reward related brain activity.
Food reward related brain activity | 12 weeks
  Difference in change between the groups. Measured using neurocognitive tests and fMRI.
  Neurocognitive functioning will be measured using CANTAB (a combination of different digital tests) to assess response time in seconds and quality of delivered results. fMRI assesses food-reward related brain activity
Tissue metabolism (subcutaneous visceral adipose tissue, skeletal muscle tissue) | 12 weeks
  Difference in change between the groups regarding receptor expression and metabolic changes in different pathways (lipolysis, insulin signalling etc)
Microbiome composition and functionality | 12 weeks
  Difference in change between the groups. Measured using 16S-RNA sequencing and faecal analysis of substrates of saccharolytic and proteolytic fermentation.
Gastrointestinal side-effects of dietary supplement | 12 weeks
  Difference in change between the groups. Measured by gastrointestinal symptom rating scale and questionnaires on general wellbeing.
  Gastro-intestinal symptom rating scale: 15 questions on 7-point Likert scale (1 = strongly disagree; 7 = strongly agree)
Stool consistency | 12 weeks
  Difference in change between the groups. Measured by bristol stool scale (7-point scale (1 = solid feces, 7 = severe diarrhoea)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof.Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blaak EE. Current metabolic perspective on malnutrition in obesity: towards more subgroup-based nutritional approaches? Proc Nutr Soc. 2020 Aug;79(3):331-337. doi: 10.1017/S0029665120000117. Epub 2020 Mar 3. PMID 32122428
- [Background] Blaak EE, Canfora EE, Theis S, Frost G, Groen AK, Mithieux G, Nauta A, Scott K, Stahl B, van Harsselaar J, van Tol R, Vaughan EE, Verbeke K. Short chain fatty acids in human gut and metabolic health. Benef Microbes. 2020 Sep 1;11(5):411-455. doi: 10.3920/BM2020.0057. Epub 2020 Aug 31. PMID 32865024
- [Background] Canfora EE, Jocken JW, Blaak EE. Short-chain fatty acids in control of body weight and insulin sensitivity. Nat Rev Endocrinol. 2015 Oct;11(10):577-91. doi: 10.1038/nrendo.2015.128. Epub 2015 Aug 11. PMID 26260141
- [Background] Canfora EE, Meex RCR, Venema K, Blaak EE. Gut microbial metabolites in obesity, NAFLD and T2DM. Nat Rev Endocrinol. 2019 May;15(5):261-273. doi: 10.1038/s41574-019-0156-z. PMID 30670819
- [Background] Canfora EE, van der Beek CM, Jocken JWE, Goossens GH, Holst JJ, Olde Damink SWM, Lenaerts K, Dejong CHC, Blaak EE. Colonic infusions of short-chain fatty acid mixtures promote energy metabolism in overweight/obese men: a randomized crossover trial. Sci Rep. 2017 May 24;7(1):2360. doi: 10.1038/s41598-017-02546-x. PMID 28539646